CLINICAL TRIAL: NCT00711022
Title: An Open, Prospective, Multicenter Study to Evaluate the Outcome of ASTRA TECH Implant System, OsseoSpeed™ Implants, in Patients With Totally Edentulous Maxillas and Poor Bone Quality and Quantity in an Immediate Loading Protocol.
Brief Title: Study on ASTRA TECH Implant System, OsseoSpeed™ Implants in Patients Missing All Teeth in the Upper Jaw, Restored With Provisional Teeth Within 24 Hours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA-OSS-0008
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-05

CONDITIONS: Jaw, Edentulous
Keywords: Jaw, Edentulous (maxilla, with poor bone quality and quantity)
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OsseoSpeed (Experimental)
  Interventions: Device: ASTRA TECH Implant System, OsseoSpeed™, all dimensions.

INTERVENTIONS:
Device: ASTRA TECH Implant System, OsseoSpeed™, all dimensions.

SUMMARY:
The purpose of the study is to evaluate ASTRA TECH Implant System, OsseoSpeed™ implants, in patients with totally edentulous upper jaws and poor bone quality and quantity, when provisional artificial teeth are attached within 24 hours. The primary objective is to investigate implant survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Aged 20 years and over
* History of totally edentulous maxilla of at least three months
* Radiographic finding indicating bone quality class 3 or 4 (Lekholm and Zarb) in the maxilla
* Radiographic finding indicating bone quantity class C, D or E (Lekholm and Zarb) in the maxilla
* Presence of natural teeth, partial prosthesis and/or implants in the mandible, within positions 35-45 (according to the FDI digit system)
* Deemed by the investigator as likely to present an initially stable implant situation suitable for immediate loading.

Exclusion Criteria:

* Unlikely to be able to comply with study procedures, as judged by the investigator
* Uncontrolled pathologic processes in the oral cavity
* Known or suspected current malignancy
* History of radiation in the head and neck region
* History of chemotherapy within 5 years prior to surgery
* Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
* Uncontrolled Diabetes Mellitus
* Corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
* History of bone augmentation in the maxilla within 6 months prior to surgery
* Known pregnancy at time of enrolment
* Present alcohol and/or drug abuse
* Current use of tobacco or history of tobacco use within 6 months prior to surgery
* Need for interpreter

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Toljanic, Prof., Principal Investigator — University of Chicago
Locations (2):
- The University of Chicago, MC-2108, Chicago, Illinois, United States
- Uppsala University Hospital, Dept. of Surgical Sciences, Oral and Maxillofacial Surgery, Faculty of Medicine, Uppsala, Sweden

REFERENCES:
- [Result] Toljanic JA, Baer RA, Ekstrand K, Thor A. Implant rehabilitation of the atrophic edentulous maxilla including immediate fixed provisional restoration without the use of bone grafting: a review of 1-year outcome data from a long-term prospective clinical trial. Int J Oral Maxillofac Implants. 2009 May-Jun;24(3):518-26. PMID 19587876
- [Result] Erkapers M, Ekstrand K, Baer RA, Toljanic JA, Thor A. Patient satisfaction following dental implant treatment with immediate loading in the edentulous atrophic maxilla. Int J Oral Maxillofac Implants. 2011 Mar-Apr;26(2):356-64. PMID 21483889
- [Result] Thor A, Ekstrand K, Baer RA, Toljanic JA. Three-year follow-up of immediately loaded implants in the edentulous atrophic maxilla: a study in patients with poor bone quantity and quality. Int J Oral Maxillofac Implants. 2014 May-Jun;29(3):642-9. doi: 10.11607/jomi.3163. PMID 24818203
- [Derived] Erkapers M, Segerstrom S, Ekstrand K, Baer RA, Toljanic JA, Thor A. The influence of immediately loaded implant treatment in the atrophic edentulous maxilla on oral health related quality of life of edentulous patients: 3-year results of a prospective study. Head Face Med. 2017 Nov 10;13(1):21. doi: 10.1186/s13005-017-0154-0. PMID 29126426

RESULTS

PARTICIPANT FLOW:
Groups:
- OsseoSpeed: ASTRA TECH Implant System, OsseoSpeed™, all dimensions.
Period: Overall Study
Arm/Group | OsseoSpeed
Started | 51
Completed | 40
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival Rate
Description: An implant that has failed to osseointegrate, lost its osseointegration or fractured was considered a failure effective from the date of removal. The survival rate for individual implants was analyzed at each visit. Cumulative implant survival rate was calculated using Kaplan-Meier life-table estimation and reported as percentage of survived implants.
Time Frame: At 5-year follow-up
Population: Per protocol analysis presented, this includes implants loaded within 24 hours from implant placement (306 implants in 51 subjects), of these 20 implants failed during the 5 year follow-up period.
Measure: Number; unit: percentage of implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed
Number analyzed (Participants) | 51
Number analyzed (Implants) | 306
percentage of implants | 93.10

ADVERSE EVENTS:
Arm/Group | OsseoSpeed
Serious Adverse Events (participants affected / at risk) | 5/51
Other Adverse Events (participants affected / at risk) | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OsseoSpeed (N=51)
Obstructed small intestine (Gastrointestinal disorders) | 1
Stroke (Vascular disorders) | 1
Cerebral vascular accident (Vascular disorders) | 1
Rectal issue (Gastrointestinal disorders) | 1
Drug related reaction (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less